CLINICAL TRIAL: NCT01957566
Title: The Utility of Amplified Pretracheal Stethoscope in Detecting Ventilatory Abnormalities During Propofol Sedation of Non Intubated Children: a Validation Study
Brief Title: The Utility of Pretracheal Stethoscope in Detecting Respiratory Abnormalities in Sedated Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HSC 2012-0259
Record Dates: First submitted 2013-01-17; First posted 2013-10-08 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Sedation
Keywords: propofol sedation; children; procedure sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APS (Experimental)
  Interventions: Procedure: APS

INTERVENTIONS:
Procedure: APS

SUMMARY:
The purpose of the study is to validate the diagnostic performance of the amplified pretracheal stethoscope (APS) to detect sedation-related adverse acute respiratory events in propofol sedated nonintubated children. To determine the sensitivity/specificity and positive/negative predictive value of the APS in detecting sedation-related adverse acute respiratory events in propofol sedated nonintubated children.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2 years to 18 years of age undergoing induction and maintenance of propofol sedation at the American Family Children's Hospital (AFCH) Pediatric Sedation Clinic
* American Society of Anesthesiology score (ASA) of 1-2

Exclusion Criteria:

* ASA scoring > 3
* Oxygen requirement and cardiorespiratory instability
* Allergy to propofol or its components
* Patients requiring propofol sedation outside the AFCH Pediatric Sedation Clinic

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
An auscultation of a stridor score greater than or equal to 2 will be defined as a sedation-related adverse acute respiratory event | Day 1 of propofol sedation.
A stridor score of less than 2 will be defined as not sedation-related event. | Day 1 of sedation.

SECONDARY OUTCOMES:
The positive predictive value and negative predictive value of the APS for predicting airway obstruction. | Day 1 of propofol sedation.
  A subject will be considered as evaluable for the sensitivity/specificity evaluation if (1) all inclusion criteria are met, (2) presedation phase is completed, and (3) the sedation induction and maintenance phase is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Boriosi, MD, Principal Investigator — UW Madison
Locations (1):
- American Family Children's Hospital (AFCH), Madison, Wisconsin, United States